CLINICAL TRIAL: NCT02244320
Title: Observational Study in Patients With Functional BPH (Benign Prostatic Hyperplasia) Symptoms Who Switched From Phytotherapy to ALNA® (Tamsulosin)
Brief Title: Observational Study in Patients With Functional Benign Prostatic Hyperplasia Symptoms Who Switched From Phytotherapy to ALNA® (Tamsulosin)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 527.38
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- functional BPH: patients with functional BPH who switched from phytotherapy to ALNA®
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Tamsulosin
  Other Names: ALNA®

SUMMARY:
The objective of the observational study were to investigate the switch from phytotherapy to ALNA® after at least 4 weeks of phytotherapy and still presented with a symptom sum score of ≥ 8 points (International Prostate Symptom Score (IPSS))

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from BPH symptoms
* Preceding treatment with a phytotherapeutic for at least 4 weeks
* IPSS sum score ≥ 8 points prior to treatment start with ALNA®
* Indication for a switch to treatment with ALNA® for a minimum period of 2 months

Exclusion Criteria:

* Patients fulfilling one of the general or specific contraindications listed in the ALNA® Summary of Product Characteristic, particularly patients with known hypersensitivities against tamsulosin hydrochloride or any other ingredient of the product, orthostatic dysregulation or severe liver insufficiency
* Patients receiving ALNA® within the 4 weeks prior to the start of the present observational study

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with functional BPH symptoms recruited at urologist offices
Sampling Method: Non-Probability Sample
Enrollment: 4150 (Actual)
Dates: Start 2002-09; Primary Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Change in IPSS sum score | Day 1, 2 months
Change in Quality-of-Life Index (QoL) rated on a 7-point scale | Day 1, 2 months

SECONDARY OUTCOMES:
Change in sexual satisfaction rated on a 4-point scale | Day 1, 2 months
Change in maximum urinary flow rate (ml/sec) | Day 1, 2 months
Change in residual urine volume (ml) | Day 1, 2 months
Patient's global assessment of the preceding phytotherapy on a 3-point scale | Day 1
Patient's global assessment of the therapy with ALNA® on a 3-point scale | after 2 months
Efficacy assessment of the preceding phytotherapy by physician rated on 4-point scale | Day 1
Efficacy assessment of the therapy with ALNA® by physician rated on 4-point scale | after 2 months
Tolerability assessment of the preceding phytotherapy by physician rated on 4-point scale | Day 1
Tolerability assessment of the therapy with ALNA® by physician rated on 4-point scale | after 2 months
Number of patients with adverse drug reactions (ADR) | up to 2 months